CLINICAL TRIAL: NCT02764918
Title: Field Studies of Cryptosporidiosis and Enteropathogens in Bangladesh
Brief Title: Cryptosporidiosis and Enteropathogens in Bangladesh
Status: Active, not recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, William Petri, MD, PhD, Division Chief, Infectious Disease, University of Virginia
Other Study IDs: PR13092; R01AI043596 (NIH)
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cryptosporidiosis
MeSH Terms: conditions — Cryptosporidiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children: n=150
- Mothers: n=150

SUMMARY:
The purpose of this study is to explore the role of anti-parasite antibody in protection of children from the parasitic infection cryptosporidiosis. This work has the promise of identifying immune pathways important for protection from parasitic infections of the gut, and will help with designing a vaccine to prevent this infection estimated to cause, from diarrhea and malnutrition, an overall burden of 12 million disability-adjusted life-years in children.

ELIGIBILITY:
Inclusion Criteria:

* Mother willing to sign informed consent form.
* Healthy infant
* No obvious congenital abnormalities or birth defects.
* Stable household with no plans to leave the area for the next one year.

Exclusion Criteria:

* Parents are not willing to have child's blood drawn.
* Parents are planning to enroll child into another interventional clinical study during the time period of this trial that could affect the outcomes of this study.
* Mother not willing to have blood drawn and breast milk extracted.
* Parents not willing to have field research assistant in home two times per week.
* History of seizures or other apparent neurologic disorders.
* Infant has any sibling currently or previously enrolled in this study, including a twin.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mother-child pairs from the Mirpur Neighborhood of Dhaka, Bangladesh
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Functional characterization of anti-Cryptosporidium antibodies associated with protection | Birth until 4 years
  Measure antibody isotype and subclass, mucosal (stool) vs systemic (plasma), complement fixation and opsonophagocytosis using bead-based multiplex immunoassays.

SECONDARY OUTCOMES:
In depth characterization of Cryptosporidium antigens recognized by the child humoral immune response | Birth until 4 years.
  Utilize this longitudinal study of children and a Cryptosporidium protein microarray to probe plasma for the breadth of antigens recognized as well as the specific antigens to which children respond as they develop protective immunity.
Polymerase chain reaction (PCR) testing for diarrheal pathogens during acute infection | Birth to 4 years old
  To be conducted on children's acute and convalescent stool during diarrheal episodes.
Determine the role of circulating T follicular helper (cTfh) cells in induction of antibody response | Through collection of blood specimens on day 0, 14 and 28 during acute infection.
  Use Activation Induced Marker (AIM) assays to test parasite infection-dependent changes in the activation, frequency, and immunophenotype of circulating Tfh cells.
Determination of maternal humoral response and impact on child infection/immunity | On enrollment (all) and 4 months (breast milk only).
  Collect mother blood, stool and breast milk on enrollment. Collect second breast milk at 4 months.
Surveillance polymerase chain reaction (PCR) testing for diarrheal pathogens | Birth until 4 years.
  To be conducted on child non diarrheal stool collected twice monthly.
Determine child anthropometric measures | Every 6 months until 4 years
  Collect height, weight, mid-upper arm circumference.
Socioeconomic status questionnaire | At enrollment
  To be conducted on mothers.
Household sanitation questionnaire | At enrollment
  To be conducted on mothers.

CONTACTS AND LOCATIONS:
Locations (1):
- The International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilchrist CA, Cotton JA, Burkey C, Arju T, Gilmartin A, Lin Y, Ahmed E, Steiner K, Alam M, Ahmed S, Robinson G, Zaman SU, Kabir M, Sanders M, Chalmers RM, Ahmed T, Ma JZ, Haque R, Faruque ASG, Berriman M, Petri WA. Genetic Diversity of Cryptosporidium hominis in a Bangladeshi Community as Revealed by Whole-Genome Sequencing. J Infect Dis. 2018 Jun 20;218(2):259-264. doi: 10.1093/infdis/jiy121. PMID 29514308
- [Background] Steiner KL, Ahmed S, Gilchrist CA, Burkey C, Cook H, Ma JZ, Korpe PS, Ahmed E, Alam M, Kabir M, Tofail F, Ahmed T, Haque R, Petri WA Jr, Faruque ASG. Species of Cryptosporidia Causing Subclinical Infection Associated With Growth Faltering in Rural and Urban Bangladesh: A Birth Cohort Study. Clin Infect Dis. 2018 Oct 15;67(9):1347-1355. doi: 10.1093/cid/ciy310. PMID 29897482
- [Background] Steiner KL, Kabir M, Priest JW, Hossain B, Gilchrist CA, Cook H, Ma JZ, Korpe PS, Ahmed T, Faruque ASG, Haque R, Petri WA. Fecal Immunoglobulin A Against a Sporozoite Antigen at 12 Months Is Associated With Delayed Time to Subsequent Cryptosporidiosis in Urban Bangladesh: A Prospective Cohort Study. Clin Infect Dis. 2020 Jan 2;70(2):323-326. doi: 10.1093/cid/ciz430. PMID 31131855
- [Background] Donowitz JR, Drew J, Taniuchi M, Platts-Mills JA, Alam M, Ferdous T, Shama T, Islam MO, Kabir M, Nayak U, Haque R, Petri WA. Diarrheal Pathogens Associated With Growth and Neurodevelopment. Clin Infect Dis. 2021 Aug 2;73(3):e683-e691. doi: 10.1093/cid/ciaa1938. PMID 33399861
- [Background] Donowitz JR, Pu Z, Lin Y, Alam M, Ferdous T, Shama T, Taniuchi M, Islam MO, Kabir M, Nayak U, Faruque ASG, Haque R, Ma JZ, Petri WA Jr. Small Intestine Bacterial Overgrowth in Bangladeshi Infants Is Associated With Growth Stunting in a Longitudinal Cohort. Am J Gastroenterol. 2022 Jan 1;117(1):167-175. doi: 10.14309/ajg.0000000000001535. PMID 34693912
- [Background] Kabir M, Alam M, Nayak U, Arju T, Hossain B, Tarannum R, Khatun A, White JA, Ma JZ, Haque R, Petri WA Jr, Gilchrist CA. Nonsterile immunity to cryptosporidiosis in infants is associated with mucosal IgA against the sporozoite and protection from malnutrition. PLoS Pathog. 2021 Jun 28;17(6):e1009445. doi: 10.1371/journal.ppat.1009445. eCollection 2021 Jun. PMID 34181697
- [Background] Carey MA, Medlock GL, Alam M, Kabir M, Uddin MJ, Nayak U, Papin J, Faruque ASG, Haque R, Petri WA, Gilchrist CA. Megasphaera in the Stool Microbiota Is Negatively Associated With Diarrheal Cryptosporidiosis. Clin Infect Dis. 2021 Sep 15;73(6):e1242-e1251. doi: 10.1093/cid/ciab207. PMID 33684930
- [Background] Gilchrist CA, Campo JJ, Pablo JV, Ma JZ, Teng A, Oberai A, Shandling AD, Alam M, Kabir M, Faruque ASG, Haque R, Petri WA Jr. Specific Cryptosporidium antigens associate with reinfection immunity and protection from cryptosporidiosis. J Clin Invest. 2023 Aug 15;133(16):e166814. doi: 10.1172/JCI166814. PMID 37347553
- [Derived] Gilchrist CA, Petri WAO, Hossain B, Kabir M, So HH, Moreau GB, Nayak U, Ma JZ, Noor Z, Faruque ASG, Alam M, Haque R, Petri WA Jr. Decrease in Incidence of Diarrhea Due to Cryptosporidium in Bangladeshi Children Is Associated With an Increase in Anti-Cryptosporidium Antibody Avidity. J Infect Dis. 2025 Sep 15;232(3):e362-e371. doi: 10.1093/infdis/jiaf253. PMID 40488529
- [Derived] Carey M, Arju T, Cotton JA, Alam M, Kabir M, Faruque ASG, Haque R, Petri WA Jr, Gilchrist CA. Genomic Heterogeneity of Cryptosporidium parvum Isolates From Children in Bangladesh: Implications for Parasite Biology and Human Infection. J Infect Dis. 2023 Nov 2;228(9):1292-1298. doi: 10.1093/infdis/jiad257. PMID 37832036